CLINICAL TRIAL: NCT04712162
Title: The Quality of Recovery After General Anesthesia With Desflurane and Sevoflurane in Endoscopic Ureteral Lithotripsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gia Dinh People Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81/CN-HĐĐĐ
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D: maintain anesthesia with desflurane (Other): D: maintain anesthesia with Suprane® (Desflurane) at 6%. Volatile concentration was titrated according to end-tidal MAC to maintain 0.7-1.3 MAC using end-tidal monitor of Dräger Primus anesthesia machine.
  Interventions: Other: Other
- S: maintain anesthesia with sevoflurane. (Other): S: maintain anesthesia with Sevorane® (Sevoflurane) at 2%. Volatile concentration was titrated according to end-tidal MAC to maintain 0.7-1.3 MAC using end-tidal monitor of Dräger Primus anesthesia machine.
  Interventions: Other: Other

INTERVENTIONS:
Other: Other — Compare time to awakening and quality of recovery after general anesthesia between two groups.

SUMMARY:
The good quality of recovery after general anesthesia is one of goals for short procedures and ambulatory surgeries. The study's objective was to compare the quality of recovery after general anesthesia with desflurane and sevoflurane with laryngeal mask airway for endoscopic ureteral lithotripsy.

DETAILED DESCRIPTION:
This is a randomized controlled trial. There were 60 cases of endoscopic ureteral lithotripsy under general anesthesia with laryngeal mask airway were enrolled. All cases were randomly divided into two group (desflurane or sevoflurane). Each group had 30 cases. Primary outcome was time to awakening. Secondary outcomes were time to wash-out of volatile anesthetics, time to extubation, irritation after awakening, and modified Aldrete score.

Statistical analysis was performed by using Kaplan-Meieir curve and log-rank test for time to adequate depth of anesthesia and time to awakening; t-test for time to wash-out of volatile anesthetics; chi-square test for depth of anesthesia by PRST score, irritation after awakening and Aldrete score; Fisher test for adverse effects of volatile anesthetics.

The research was approved by Gia Dinh People Hospital ethics committee

ELIGIBILITY:
Inclusion Criteria:

* All eligible subjects who underwent endoscopic ureteral lithotripsy under general anesthesia
* ASA I and II

Exclusion Criteria:

* Contraindication to laryngeal mask airway.
* Indication for conversion to tracheal intubation during surgery.
* History of malignant hyperthermia.
* Pregnancy.
* Obese (BMI >25 kg/m2).
* Substances abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Time to awakening | After stopping volatile anesthetics to patient awakening, up to 30 minutes.
  Time required for awakening

SECONDARY OUTCOMES:
Time to wash-out of volatile anesthetics | After stopping volatile anesthetics to complete wash-out of volatile anesthetics, up to 30 minutes
  Time required for washing out volatile anesthetics
Time to extubation | After stopping volatile anesthetics to readiness for extubation, up to 30 minutes
  Time required for successful extubation.
Irritation after awakening | After awakening to eligible discharge, up to 2 hours.
  Aono score >2
Adverse effects of volatile anesthetics | After providing volatile anesthetics until they were stopped, up to 90 minutes
  Hypotension, cough, nausea and vomitting.

CONTACTS AND LOCATIONS:
Overall Officials: Thanh T. Nguyen, PhD, Study Chair — Gia Dinh People Hospital
Locations (1):
- Anesthesiology Department of Gia Dinh People Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code

REFERENCES:
- [Background] Bruhn J, Bouillon TW, Shafer SL. Bispectral index (BIS) and burst suppression: revealing a part of the BIS algorithm. J Clin Monit Comput. 2000;16(8):593-6. doi: 10.1023/A:1012216600170. PMID 12580235
- [Background] Drover DR, Lemmens HJ, Pierce ET, Plourde G, Loyd G, Ornstein E, Prichep LS, Chabot RJ, Gugino L. Patient State Index: titration of delivery and recovery from propofol, alfentanil, and nitrous oxide anesthesia. Anesthesiology. 2002 Jul;97(1):82-9. doi: 10.1097/00000542-200207000-00012. PMID 12131107
- [Background] Eger EI 2nd, Saidman LJ, Brandstater B. Minimum alveolar anesthetic concentration: a standard of anesthetic potency. Anesthesiology. 1965 Nov-Dec;26(6):756-63. doi: 10.1097/00000542-196511000-00010. No abstract available. PMID 5844267
- [Background] Katoh T, Ikeda K. The effects of fentanyl on sevoflurane requirements for loss of consciousness and skin incision. Anesthesiology. 1998 Jan;88(1):18-24. doi: 10.1097/00000542-199801000-00006. PMID 9447851
- [Background] Katoh T, Kobayashi S, Suzuki A, Iwamoto T, Bito H, Ikeda K. The effect of fentanyl on sevoflurane requirements for somatic and sympathetic responses to surgical incision. Anesthesiology. 1999 Feb;90(2):398-405. doi: 10.1097/00000542-199902000-00012. PMID 9952144
- [Background] Rampil IJ, Lockhart SH, Zwass MS, Peterson N, Yasuda N, Eger EI 2nd, Weiskopf RB, Damask MC. Clinical characteristics of desflurane in surgical patients: minimum alveolar concentration. Anesthesiology. 1991 Mar;74(3):429-33. doi: 10.1097/00000542-199103000-00007. PMID 2001020
- [Background] Whitlock EL, Villafranca AJ, Lin N, Palanca BJ, Jacobsohn E, Finkel KJ, Zhang L, Burnside BA, Kaiser HA, Evers AS, Avidan MS. Relationship between bispectral index values and volatile anesthetic concentrations during the maintenance phase of anesthesia in the B-Unaware trial. Anesthesiology. 2011 Dec;115(6):1209-18. doi: 10.1097/ALN.0b013e3182395dcb. PMID 22037642
- [Result] Aldrete JA. Post-anesthetic recovery score. J Am Coll Surg. 2007 Nov;205(5):e3-4; author reply e4-5. doi: 10.1016/j.jamcollsurg.2007.07.034. No abstract available. PMID 17964430
- [Result] Aldrete JA, Kroulik D. A postanesthetic recovery score. Anesth Analg. 1970 Nov-Dec;49(6):924-34. No abstract available. PMID 5534693
- [Result] Choi GJ, Baek CW, Kang H, Park YH, Yang SY, Shin HY, Jung YH, Woo YC, Lee UL. Emergence agitation after orthognathic surgery: a randomised controlled comparison between sevoflurane and desflurane. Acta Anaesthesiol Scand. 2015 Feb;59(2):224-31. doi: 10.1111/aas.12435. Epub 2014 Nov 14. PMID 25395384
- [Result] De Oliveira GS Jr, Fitzgerald PC, Ahmad S, Marcus RJ, McCarthy RJ. Desflurane/fentanyl compared with sevoflurane/fentanyl on awakening and quality of recovery in outpatient surgery using a laryngeal mask airway: a randomized, double-blinded controlled trial. J Clin Anesth. 2013 Dec;25(8):651-8. doi: 10.1016/j.jclinane.2013.07.006. Epub 2013 Oct 4. PMID 24095885
- [Result] Dogru K, Yildiz K, Madenoglu H, Boyaci A. Early recovery properties of sevoflurane and desflurane in patients undergoing total hip replacement surgery. Curr Ther Res Clin Exp. 2003 May;64(5):301-9. doi: 10.1016/S0011-393X(03)00086-9. PMID 24944378
- [Result] Green MS, Green P, Neubert L, Voralu K, Saththasivam P, Mychaskiw G. Recovery following desflurane versus sevoflurane anesthesia for outpatient urologic surgery in elderly females. Anesth Pain Med. 2015 Feb 1;5(1):e22271. doi: 10.5812/aapm.22271. eCollection 2015 Feb. PMID 25789236
- [Result] Kaur A, Jain AK, Sehgal R, Sood J. Hemodynamics and early recovery characteristics of desflurane versus sevoflurane in bariatric surgery. J Anaesthesiol Clin Pharmacol. 2013 Jan;29(1):36-40. doi: 10.4103/0970-9185.105792. PMID 23493107
- [Result] La Colla L, Albertin A, La Colla G, Mangano A. Faster wash-out and recovery for desflurane vs sevoflurane in morbidly obese patients when no premedication is used. Br J Anaesth. 2007 Sep;99(3):353-8. doi: 10.1093/bja/aem197. Epub 2007 Jul 9. PMID 17621601
- [Result] Mahmoud NA, Rose DJ, Laurence AS. Desflurane or sevoflurane for gynaecological day-case anaesthesia with spontaneous respiration? Anaesthesia. 2001 Feb;56(2):171-4. doi: 10.1046/j.1365-2044.2001.01528.x. PMID 11167479
- [Result] Mikuni I, Harada S, Yakushiji R, Iwasaki H. Effects of changing from sevoflurane to desflurane on the recovery profile after sevoflurane induction: a randomized controlled study. Can J Anaesth. 2016 Mar;63(3):290-7. doi: 10.1007/s12630-015-0514-9. Epub 2015 Oct 20. PMID 26487303
- [Result] Saros GB, Doolke A, Anderson RE, Jakobsson JG. Desflurane vs. sevoflurane as the main inhaled anaesthetic for spontaneous breathing via a laryngeal mask for varicose vein day surgery: a prospective randomized study. Acta Anaesthesiol Scand. 2006 May;50(5):549-52. doi: 10.1111/j.1399-6576.2006.001022.x. PMID 16643222
- [Result] Smajic J, Praso M, Hodzic M, Hodzic S, Srabovic-Okanovic A, Smajic N, Djonlagic Z. Assessment of depth of anesthesia: PRST score versus bispectral index. Med Arh. 2011;65(4):216-20. doi: 10.5455/medarh.2011.65.216-220. PMID 21950227
- [Result] Werner JG, Castellon-Larios K, Thongrong C, Knudsen BE, Lowery DS, Antor MA, Bergese SD. Desflurane Allows for a Faster Emergence When Compared to Sevoflurane without Affecting the Baseline Cognitive Recovery Time. Front Med (Lausanne). 2015 Oct 28;2:75. doi: 10.3389/fmed.2015.00075. eCollection 2015. PMID 26579522
- [Result] Wissing H, Kuhn I, Rietbrock S, Fuhr U. Pharmacokinetics of inhaled anaesthetics in a clinical setting: comparison of desflurane, isoflurane and sevoflurane. Br J Anaesth. 2000 Apr;84(4):443-9. doi: 10.1093/oxfordjournals.bja.a013467. PMID 10823093